CLINICAL TRIAL: NCT04213222
Title: A Radiomics Approach to Predict the Effect of Bevacizumab Plus Chemotherapy in Patients With Liver Metastases of Colorectal Cancer: A Prospective Multi-Centers Trial
Brief Title: Radiomics Assess of Bevacizumab Plus Chemo in Colorectal Cancer Liver Metastases
Acronym: ROBOT
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 20181113
Record Dates: First submitted 2019-12-25; First posted 2019-12-30 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Colon Cancer; Rectal Cancer; Liver Metastases
Keywords: colorectal cancer; liver metastasis; bevacizumab
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms; Colorectal Neoplasms | interventions — Bevacizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Bevacizumab — bevacizumab combined with chemotherapy

SUMMARY:
Colorectal carcinoma with liver metastasis is one of the major problems bothering physicians worldwide. Bevacizumab combined with chemotherapy is the standard treatment recommended by several guidelines. Despite the high cost, a certain portion of patients couldn't benefit from this therapy. This study is aiming to find out the specific type of patients who would respond to bevacizumab by Radiomics approach, and evaluate the prediction value of this imaging model with clinical and genetic factors.

ELIGIBILITY:
Inclusion Criteria:

1. Colorectal carcinoma confirmed by pathological result.
2. Liver metastasis confirmed by imaging studies.
3. Treatment of bevacizumab combined with chemotherapy chosen by MDT team.
4. ECOG: 0-2.
5. Normal laboratory studies including liver\renal\bone marrow functions.
6. Expected lifespan more than 3 months.

Exclusion Criteria:

1. Previous treatment of colorectal cancer with liver metastasis.
2. Diagnosed with other malignancies.
3. Couldn't finish the trial due to several reasons such as allergy to chemotherapy drugs\pregnancy or lactation\chronic heart disease\unable to sustain further treatment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of colorectal carcinoma with liver metastasis
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-10 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
estimated ORR | 6-8 weeks

SECONDARY OUTCOMES:
estimated PFS | 3 years
estimated OS | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided